CLINICAL TRIAL: NCT06874621
Title: VY7523-102: A Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Multiple Ascending Intravenous Doses of VY7523 in Participants With Early Alzheimer's Disease
Brief Title: VY7523-102: Randomized, Placebo-Controlled, Double-Blind, Multiple Ascending Dose Study in Participants With Early Alzheimer's Disease
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Voyager Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VY7523-102
Record Dates: First submitted 2025-03-04; First posted 2025-03-13 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer's Disease (AD)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 active (Experimental): Low dose VY7523
  Interventions: Drug: VY7523
- Cohort 1 placebo (Placebo Comparator): VY7523 matching placebo for Cohort 1 active dose
  Interventions: Drug: Placebo Comparator
- Cohort 2 active (Experimental): mid dose VY7523
  Interventions: Drug: VY7523
- Cohort 2 placebo (Placebo Comparator): VY7523 matching placebo for Cohort 2 active dose
  Interventions: Drug: Placebo Comparator
- Cohort 3 active (Experimental): high dose VY7523
  Interventions: Drug: VY7523
- Cohort 3 placebo (Placebo Comparator): VY7523 matching placebo for Cohort 3 active dose
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: VY7523 — VY7523 is a recombinant humanized immunoglobulin gamma 4 (IgG4) monoclonal antibody targeting human pathological tau
  Arms: Cohort 1 active; Cohort 2 active; Cohort 3 active
Drug: Placebo Comparator — Matching placebo to VY7523
  Arms: Cohort 1 placebo; Cohort 2 placebo; Cohort 3 placebo

SUMMARY:
This study is to be conducted in participants with early Alzheimer's Disease to test VY7523, a new drug being researched for treatment of Alzheimer's Disease. This study will look at how safe the drug is and how it works in the brain. It was first tested in normal, healthy participants who volunteered to participate. The study will look at three different dose levels, starting with the lowest dose first and moving to higher doses and more participants after safety has been reviewed by doctors and researchers. Some patients will receive drug while others will receive placebo. This will help to better compare how the drug works between participants receiving drug and placebo. The study will last up to 6 months for the lower dose groups and 12 months for the highest dose group.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of early AD, defined as:

   1. Meet the NIA-AA core clinical criteria for MCI due to AD or mild AD.
   2. Mini Mental State Examination (MMSE) score between 18 and 30, inclusive, at Screening (Cohort 1 and 2) and score between 22 and 30, inclusive, at Screening (Cohort 3).
   3. Report a history of subjective memory decline with gradual onset and slow progression over at least the last 6 months before Screening; must be corroborated by an informant/caregiver.
   4. CDR Memory Box score ≥0.5 CDR global score of 0.5 for MCI due to AD or 0.5 or 1 for mild AD.
2. Evidence of pathology consistent with AD diagnosis:

   1. For Cohort 1 and Cohort 2 only, by documented historical amyloid PET showing imaging agent uptake into the brain conducted within 24 months before screening OR elevated plasma pTau217/np-Tau217 ratio within the Screening Period.
   2. For Cohort 3 only, evidence of pathology consistent with AD diagnosis by both:

      * Evidence of Tau PET imaging agent uptake into the brain by central read AND
      * Evidence of positive brain amyloid pathology as indicated by one of the following:

   <!-- -->

   1. Documented historical amyloid PET showing imaging agent uptake into the brain conducted within 24 months before screening OR
   2. CSF beta amyloid and tau levels consistent with AD diagnosis within the Screening Period.
3. Body mass index (BMI) ≥18 and ≤35 kg/m2 at Screening.
4. Apart from the clinical diagnosis of early AD, participant must be in good health, based on medical history and screening assessments.
5. If participant is receiving an approved symptomatic AD treatment such as but not limited to acetylcholinesterase inhibitor (AChEIs), memantine, rivastigmine, galantamine and tacrine for AD, participant must be on a stable dose for at least 8 weeks prior to Screening.

   1. Treatment-naive participants for AD can be entered into the study.
   2. Unless otherwise stated, participants must have been on stable doses of all other (non-AD-related) permitted concomitant medications for at least 4 weeks prior to Screening.
   3. Participants currently on β amyloid therapies may not be enrolled.
6. Must have an identified reliable informant/caregiver (defined as a person able to support the participant for the duration of the study e.g., spouse, sibling, close friend, who spends at least 10 hours per week with the participant) who assented to:

   1. Accompany the participant to clinic visits.
   2. Provide information to study Investigator/staff about functioning, cognitive abilities and AEs.
   3. Support participants returning for per-protocol follow-up visits and procedures.

Exclusion Criteria:

1. Any medical or neurological/neurodegenerative or psychiatric condition (other than AD) that, in the opinion of the Investigator, may be contributing cause to cognitive impairment or could confound interpretation of drug effect, affect study assessments, or affect participant's ability to participate and complete the study or lead to safety concerns.
2. History of transient ischemic attack or stroke or any unexplained loss of consciousness within 1 year prior to Screening.
3. History of seizures within 10 years prior to screening or history of epileptic syndrome (except for history of febrile seizures in childhood)
4. Lifetime history of a major psychiatric disorder including schizophrenia or bipolar disorder. History of major depressive disorder that has resulted in 2 or more hospitalizations in a lifetime.
5. Presence of a clinically significant uncontrolled medical disorder involving one or more of these major organ systems: cardiovascular (including but not limited to a QTcF of >470 ms for women and >450 ms for men and uncontrolled hypertension), respiratory, renal, gastrointestinal, immunologic, hematologic including bleeding disorder, hepatic, or endocrine.
6. Contraindications to lumbar puncture, including but not limited to coagulation or bleeding disorders, unsafe suspension of anticoagulant, infections at the injection site, spinal deformities or previous spinal surgeries that may affect safe LP performance, or conditions associated with increased intracranial pressure.
7. Contraindications to MRI scanning, including but not limited to cardiac pacemaker/defibrillator, ferromagnetic metal implants (devices other than those approved as safe for use in MRI scanners).
8. History of a malignant disease (cancer) except for resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, in situ prostate cancer with a normal posttreatment prostate-specific antigen within the last five years or other cancers in remission for at least 5 years
9. Any immunological disease which is not adequately controlled, or which requires treatment with immunoglobulins, systemic mAbs (or derivatives of mAbs), systemic immunosuppressants, or plasmapheresis during the study.
10. History of severe allergies, or history of an anaphylactic reaction (nonactive hay fever is acceptable).
11. Participation in a clinical drug trial or device within 30 days (or 5 half-lives, whichever is longer and 3 months for a biologic) of screening, unless the study blind has been broken and the participant was known to be on placebo.
12. Last administration of B-secretase and gamma-secretase inhibitors in a study within 3 months or 5 half-lives (whichever is longer) prior to screening, unless it can be documented that the participant only received placebo.
13. Current use of an approved AD disease modifying or anti-amyloid therapy (including but not limited to any mAb therapies).
14. Presence of risk for increased or uncontrolled bleeding and/or risk of bleeding that is not managed optimally and could place a participant at an increased risk for intraoperative or postoperative bleeding.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Characterization of the safety and tolerability of VY7523 in participants with early AD | Cohorts 1 and 2: up to 6 months Cohort 3: up to 12 months
  Incidence of treatment-emergent adverse events (TEAEs) and clinically significant changes from baseline

SECONDARY OUTCOMES:
To characterize the pharmacokinetics (PK) of VY7523 in serum | Cohort 1 & 2: Month 1 - 6 Cohort 3: Month 1-7, 9, 12
  • Serum VY7523 concentrations
To evaluate the ability of VY7523 to prevent the spread of pathologic tau; Cohort 3 only | Month 6, 12
  Changes from baseline in the standardized uptake value ratio (SUVR) using tau-positron emission tomography (PET)
To evaluate the immunogenicity of multiple, escalating intravenous (IV) doses of VY7523 | Cohort 1 & 2: Month 1, 3, 4, 5 & 6 Cohort 3: Month 1, 2, 6, 9, 12
  Incidence and level of treatment emergent anti-drug antibodies to VY7523
To characterize the pharmacokinetics (PK) of VY7523 in cerebrospinal fluid (CSF) concentrations following multiple IV doses | Cohort 1 & 2: Month 6 Cohort 3: Month 12
  VY7523 CSF concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Voyager Therapuetics, Inc.
Locations (23):
- United States (19):
  - VYGR Site 840018, Los Angeles, California
  - VYGR Site 840016, Orange, California
  - VYGR Site 840022, San Francisco, California
  - VYGR Site 840008, Stamford, Connecticut
  - VYGR Site 840005, Delray Beach, Florida
  - VYGR Site 840021, Fort Myers, Florida
  - VYGR Site 840010, Lady Lake, Florida
  - VYGR Site 840015, Miami, Florida
  - VYGR Site 840014, Miami, Florida
  - VYGR Site 840024, Miami, Florida
  - VYGR Site 840006, Orlando, Florida
  - VYGR Site 840003, Stuart, Florida
  - VYGR Site 840004, The Villages, Florida
  - VYGR Site 840002, Wellington, Florida
  - VYGR Site 840020, Winter Park, Florida
  - VYGR Site 840007, Decatur, Georgia
  - VYGR Site 840012, Toms River, New Jersey
  - VYGR Site 840009, Matthews, North Carolina
  - VYGR Site 840011, Plymouth Meeting, Pennsylvania
- Canada (4):
  - VYGR Site 124002, Ottawa, Ontario
  - VYGR Site 124001, Toronto, Ontario
  - VYGR Site 124003, Montreal, Quebec
  - VYGR Site 124004, Montreal, Quebec